CLINICAL TRIAL: NCT05895773
Title: Effect of Nasal and Oropharyngeal Use of Povidone Iodine and Glycyrrhizin on Ventilator-associated Respiratory Infections: A Randomized Trial
Brief Title: Oro-nasal Decontamination to Prevent Ventilator-associated Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hazem Ezzat Elsersy, assistant professor of anesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4/2023ANET2
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Povidone-Iodine; Glycyrrhizic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated using a computer program into two equal groups: the treatment group and the placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the pharmacist is aware of the randomization and preparing the study drugs. The pharmacist will encode the medication bottles and keep the code key confidential until the completion of follow-up of the last patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Nasal and oropharyngeal Povidone Iodine plus Glycyrrhizin sprays will be applied 4 times daily after tooth cleaning with a brush.
  Interventions: Drug: Povidone-Iodine
- Placebo group (Placebo Comparator): Nasal and oropharyngeal saline sprays will be applied 4 times daily after teeth cleaning with a brush.
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Povidone-Iodine — Povidone Iodine 0.5% plus glycyrrhizin acid 2.5 mg/ml as a nasal and an oropharyngeal spray (mint flavored) will be applied 4 times per day.
  Other Names: glycyrrhizic acid
  Arms: Treatment group
Drug: Saline spray — Normal saline 0.9% as a nasal and oropharyngeal spray (Mint flavored) will be applied 4 times per day.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
It has been shown that oral hygiene reduces the incidence of ventilator-associated pneumonia (VAP). The nasopharynx is considered to be an important source of contaminated micro aspiration to the lung however, the effect of nasopharyngeal decontamination on VAP has not been yet investigated. The investigators hypothesized that decontamination of oral and nasopharyngeal cavities with combined Povidone Iodine and glycyrrhizin would remarkably reduce the incidence of VAP.

DETAILED DESCRIPTION:
Infections that occur more than 48 hours after intubation are known as ventilator-associated pneumonia (VAP) and ventilator-associated tracheobronchitis (VAT). The incidence of VAP in mechanically ventilated patients ranges from 8 to 48% with a mortality rate of 24%-76%.

These infections are a serious problem that Increases the need for prolonged hospitalization, antimicrobial therapy, and rising healthcare expenses. As a result, preventing VAP and VAT is critical to improving the quality of life by reducing complications in mechanically ventilated patients.

Intubation is a mechanical procedure that Breaks the natural barrier, allowing bacteria to colonize. Microorganisms enter the lungs through the lower respiratory tract from the oropharynx, the endotracheal tube cuff leaks, or the biofilm in the endotracheal tube. The microbial flora in the oral cavities of hospitalized patients, particularly those mechanically ventilated, gradually changes; gram-positive bacteria of low virulence predominate at admission (Streptococcus spp., Actinomyces spp.) are gradually replaced by more virulent gram-negative, potentially pathogenic microbial flora. This change happens on mucosal surfaces as well as in dental plaque, which in the physiological state are populated by 200-350 different bacterial species. The nasal-oropharyngeal axis involves nasal secretions swept to the oropharynx by mucociliary clearance followed by the aspiration of infected fluid into the lower airway. Nasal-oropharyngeal axis with subsequent seeding of the lungs leads to respiratory disease. The investigators hypothesized that micro aspirates from the nasopharynx and oropharynx are substantially contributing to the development of both VAT and VAP and the decontamination of the nasal and oral cavity would greatly help in the reduction of VAP and VAT. The purpose of this study is to compare the effect of nasal and Oro-pharyngeal use of a combination of Povidone Iodine (PVI) and Glycyrrhizin (GA) [treatment group] for oral and nasal decontamination on preventing VAP and VAT with the placebo group. Another objective is to compare the effect of treatment used for oral care on oral health and the prevention of microbial colonization in the mouth with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* on mechanical ventilation less than 24 h after admission and expected to continue mechanical ventilation for more than 72h.

Exclusion Criteria:

* Exclusion criteria include immunosuppression, aspiration pneumonia, all types of pneumonia, sepsis and septic shock, tracheostomy, and pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
ventilator-associated pneumonia. | every day for 15 days
  Clinical criteria for VAP include the following: worsened or development of new infiltrates in chest radiographs, body temperature less than 35°C or more than 38.5 °C, the leukocytic count below 4000 /mm3 or more than 11000/ mm3, tracheal aspirate of sputum or purulent discharge, and the demand for a positive end-expiratory pressure by more than 20% to keep oxygen saturation above 92% or the need for an increase in the inspired oxygen fraction. Each parameter is given a score of 0, 1, or 2. A score of 6 or more confirms VAP.

SECONDARY OUTCOMES:
Beck oral assessment score. | 4,8 and 12 hours after oral hygiene.
  Examination of lips, gingiva, oral mucosa, tongue, teeth, and saliva each given 1 to 4 according to severity. a total score of 5 denotes no dysfunction while a score from 16 to 20 indicates severe dysfunction.
Mechanical ventilation length. | up to 24 weeks.
  Days spent by the patient on the ventilator.
Mortality | up to 6 months.
  Percentage of patients died from VAP.
Length of ICU stay. | up to 24 weeks.
  Number of days patients need to be discharged from ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem E Elsersy, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia University hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: access criteria will be open for researchers, all data will be released except for personal identification for patients. To request data please contact the principal investigator e-mail. hazelsersy@hotmail.com